CLINICAL TRIAL: NCT02113033
Title: VAgal Nerve Stimulation: safeGUARDing Heart Failure Patients
Acronym: VANGUARD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVNS01
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Intervention Model Description: Equilia VNS device
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated with Equilia system (Experimental): Implantation and activation of the Vagus Nerve Stimulator, nerve electrode and cardiac lead
  Interventions: Device: Equilia® Vagal Nerve Stimulation

INTERVENTIONS:
Device: Equilia® Vagal Nerve Stimulation — Vagal Nerve Stimulation synchronized with cardiac activity
  Other Names: Device used: Equilia®

SUMMARY:
The purpose of the VANGUARD study is to demonstrate the safety of Vagal Nerve Stimulation for the treatment of congestive heart failure with reduced ejection fraction, and to report secondary measures of efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Left ventricular dysfunction of ischemic or idiopathic dilated cardiomyopathy etiology, characterized by LVEF < 40%
2. Chronic heart failure with symptoms characterized by NYHA functional class II or III at the time of enrollment despite optimal drug regimen
3. Optimal drug regimen as defined in the current European guidelines
4. Sinus rhythm, with spontaneous heart rate ≥ 60bpm at the time of enrollment
5. Signed and dated informed consent

Main Exclusion Criteria:

* Patient implanted with or eligible to cardiac pacing as per current guideline
* Risk for neck surgery in the electrode zone within a year after enrollment
* Patient with right carotid artery stenosis
* Symptomatic hypotension
* History of peptic ulcer disease or upper gastrointestinal bleeding
* Asthma, severe COPD, or severe restrictive lung disease
* Advanced Diabetes Mellitus
* Recent acute myocardial infarction, coronary artery surgery or revascularization (or already planned)
* Recent cerebro-vascular event
* Significant valvulopathy
* Advanced Renal failure
* Previous heart transplant or current LVAD device therapy
* Life expectancy < 1 year for non-cardiac cause
* Patient included in another clinical study that could confound the results of this study
* Inability to understand the purpose of the study or to perform the procedures of the study
* Unavailability for scheduled follow-up
* Age of less than 18 years or under guardianship
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2016-02-22 (Actual); Study Completion 2016-09-20 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the freedom from Serious Adverse Device Effects, defined as the number of patients without SADEs. | 6 Months
  Adverse device effects will be sub-classified into device-related or procedure-related, when the adverse event has a generic cause independent from the device itself and occurs within 30 days of the implant procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Hagege, MD, PhD, Principal Investigator — HEGP - Paris, France
Locations (6):
- UCL St Luc, Brussels, Belgium
- France (3):
  - Hôpital Européen Georges Pompidou, Paris
  - CHRU Hôpital Pontchaillou, Rennes
  - CHU Rangueil, Toulouse
- Rikshospitalet, Oslo, Norway
- Dedinje Cardiovascular Institute, Belgrade, Serbia